CLINICAL TRIAL: NCT06579196
Title: Evaluation of Trabedersen (OT-101) With Pembrolizumab in Patients With Newly Diagnosed Advanced Non-Small Cell Lung Cancer and Positive PD-L1
Brief Title: Trabedersen (OT-101) With Pembrolizumab for Newly Diagnosed Advanced NSCLC and Positive PD-L1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0740-24-FB
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Newly Diagnosed; PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Trabedersen; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Participants are enrolled into the Phase I arm until the recommended phase 2 dose (RP2D) is determined. Participants who receive the RP2D in Phase I are reassigned to the Phase II arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I: Dose Finding (Experimental): Participants receive either 140, 190, or 250 mg/m2 intravenous OT-101/Trabedersen for up to 12 weeks using a 4 days on 10 days off dosing schedule. The dose level is determined according to the Bayesian optimal interval (BOIN) design with cohort size 3.
  Participants receive concurrent administration of 400 mg intravenous Pembrolizumab every 6 weeks.
  Interventions: Drug: Trabedersen; Drug: Pembrolizumab
- Arm II: Treatment (Experimental): Participants receive the recommended phase II dose of intravenous OT-101/Trabedersen (140, 190, or 250 mg/m2) until progression using a 4 days on 10 days off dosing schedule.
  Participants receive concurrent administration of 400 mg intravenous Pembrolizumab every 6 weeks.
  Interventions: Drug: Trabedersen; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Trabedersen — Trabedersen (OT-101) is a synthetic antisense oligodeoxynucleotide that specifically inhibits the production of Transforming growth factor-beta 2 (TGF-β2).
  Other Names: OT101
Drug: Pembrolizumab — Pembrolizumab is a humanized anti-programmed death (PD-1) monoclonal antibody.
  Other Names: Keytruda

SUMMARY:
The goal of this clinical trial is to: 1) evaluate the safety and recommended dose of the drug OT-101/Trabedersen when combined with Pembrolizumab and 2) determine the efficacy of the combination therapy in adults with certain types of Non-Small Cell Lung Cancer. The main question(s) it aims to answer are:

* What medical problems to participants have when taking OT101 together with Pembrolizumab?
* What is the correct dose of OT-101 to use when evaluating the safety and efficacy of the combination therapy?
* Does the combination therapy delay progression or relapse of the participant's Non-Small Cell Lung Cancer?

Participants will:

* Receive intravenous OT-101/Trabedersen for 4 days once every 2 weeks. Clinic visits are required to receive and disconnect the infusion.
* Receive intravenous Pembrolizumab once every 6 weeks.

DETAILED DESCRIPTION:
The goal of this clinical trial is to: 1) evaluate the safety and recommended dose of the drug OT-101/Trabedersen when combined with Pembrolizumab and 2) determine the efficacy of the combination therapy in adults with certain types of Non-Small Cell Lung Cancer. The main question(s) it aims to answer are:

* What medical problems to participants have when taking OT101 together with Pembrolizumab?
* What is the correct dose of OT-101 to use when evaluating the safety and efficacy of the combination therapy?
* Does the combination therapy delay progression or relapse of the participants Non-Small Cell Lung Cancer?

Participants will:

* Receive intravenous OT-101/Trabedersen for 4 days once every 2 weeks. Clinic visits are required to receive and disconnect the infusion.
* Receive intravenous Pembrolizumab once every 6 weeks.

In Phase I, dose escalation/de-escalation of OT101/Trabedersen is performed using a BOIN design to determine dose limiting toxicity (DLT) and the recommended phase 2 dose (RP2D) when combined with Pembrolizumab.

In Phase II, subjects receive the RP2D of OT101/Trabedersen together with Pembrolizumab until disease relapse, progression [as determined by immune Response Evaluation Criteria in Solid Tumours (iRECIST) criteria], or death.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Histologically/cytologically proven diagnosis of non-small cell lung cancer (NSCLC) with a PD-L1 of at least 1%
* Metastatic disease or disease not amenable for curative intent therapy
* No prior treatment for metastatic NSCLC. Early-stage disease therapy acceptable if completed at least six months prior and did not include immunotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Measurable disease by RECIST criteria
* Adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/mm3
  * Platelets ≥100,000/mm3
  * Hemoglobin >9.0 mg/dL
  * Creatinine clearance > 60 ml/min/1.73 m2 using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
  * Total serum bilirubin <1.5 X upper limit of normal (ULN) except if known to have Gilbert's syndrome, then excluded if total bilirubin >2.5 X ULN
  * Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) ≤ 2.5 x ULN; if participant has liver metastases, ≤5x ULN
* For females of childbearing potential, negative serum or urine pregnancy test ≤7 days of treatment, & agree to use effective contraceptive during treatment & 90 days after end of treatment
* Male participants must agree to use effective contraception during the trial & for 90 days after end of treatment
* Able to give informed consent

Exclusion Criteria:

* Received any systemic treatments including investigational agents within the last 28 days
* Known hypersensitivity to any of the excipients of OT101 or pembrolizumab
* Received radiotherapy within 14 days of the study intervention. Palliative radiation is allowed during the study with a 1-week washout
* Pregnant or breast-feeding women
* History of autoimmune diseases that required systemic treatment in the past 2 years with agents such as, but not limited to, corticosteroids or immunosuppressive drugs. Thyroid replacement for hypothyroidism, insulin treatment for type I diabetes or corticosteroids adrenal/pituitary insufficiency are allowed.
* Uncontrolled systemic diseases that in the opinion of the investigator may interfere with the protocol activities
* Known active second malignancy that needs treatment. Exceptions include basal cell or squamous cancers of the skin, bladder or cervical carcinoma in situ, prostate cancer on hormone therapy alone.
* Immunodeficiency diagnosis or receiving chronic steroids that exceed a dose equivalent to prednisone 10 mg daily
* Symptomatic brain metastases. Asymptomatic metastases or having received treatment for brain metastases and are off steroid therapy is acceptable.
* Known psychiatric or substance use that would interfere with the study requirements
* Inability to co-operate with the requirements of the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Phase I: Dose Finding | 18 months
  Dose Limiting toxicity (DLT) and Maximum Tolerated Dose (MTD)
Phase II: Progression-Free Survival (PFS) | 36 months
  Progression-Free Survival (PFS) defined as first therapy until the first documentation of clinical progression, relapse, or death due to any cause. Participants not experiencing an event of interest will be right-censored at last known disease status

SECONDARY OUTCOMES:
Best Overall Response | 36 months
  Best overall response, defined as the best overall response observed during the evaluation period (up to 12 weeks of treatment): CR, PR, SD, or PD,
Disease Control | 36 months
  Disease control [CR + PR + stable disease (SD)]
Duration of Response | 36 months
  Duration of response (DOR) defined as first response (CR or PR) until disease progression.
Drug Toxicity | 18 months
  Toxicity according to Common Terminology Criteria for Adverse Events (CTCAE).
Overall Survival (OS) | 48 months
  Overall survival (OS) defined as the time from the first therapy until death.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Abughanimeh, MBBS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abughanimeh O, Kaur A, El Osta B, Ganti AK. Novel targeted therapies for advanced non-small lung cancer. Semin Oncol. 2022 Jun;49(3-4):326-336. doi: 10.1053/j.seminoncol.2022.03.003. Epub 2022 Apr 1. PMID 35414419
- [Background] National Comprehensive Cancer Network. Non-small cell lung cancer. Version 2. 2024. Available at: https://www.nccn.org/professionals/physician_gls/pdf/nscl.pdf. Accessed Feb 12
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Mok TSK, Wu YL, Kudaba I, Kowalski DM, Cho BC, Turna HZ, Castro G Jr, Srimuninnimit V, Laktionov KK, Bondarenko I, Kubota K, Lubiniecki GM, Zhang J, Kush D, Lopes G; KEYNOTE-042 Investigators. Pembrolizumab versus chemotherapy for previously untreated, PD-L1-expressing, locally advanced or metastatic non-small-cell lung cancer (KEYNOTE-042): a randomised, open-label, controlled, phase 3 trial. Lancet. 2019 May 4;393(10183):1819-1830. doi: 10.1016/S0140-6736(18)32409-7. Epub 2019 Apr 4. PMID 30955977
- [Background] Herbst RS, Giaccone G, de Marinis F, Reinmuth N, Vergnenegre A, Barrios CH, Morise M, Felip E, Andric Z, Geater S, Ozguroglu M, Zou W, Sandler A, Enquist I, Komatsubara K, Deng Y, Kuriki H, Wen X, McCleland M, Mocci S, Jassem J, Spigel DR. Atezolizumab for First-Line Treatment of PD-L1-Selected Patients with NSCLC. N Engl J Med. 2020 Oct 1;383(14):1328-1339. doi: 10.1056/NEJMoa1917346. PMID 32997907
- [Background] Ozguroglu M, Kilickap S, Sezer A, Gumus M, Bondarenko I, Gogishvili M, Nechaeva M, Schenker M, Cicin I, Ho GF, Kulyaba Y, Zyuhal K, Scheusan RI, Garassino MC, He X, Kaul M, Okoye E, Li Y, Li S, Pouliot JF, Seebach F, Lowy I, Gullo G, Rietschel P. First-line cemiplimab monotherapy and continued cemiplimab beyond progression plus chemotherapy for advanced non-small-cell lung cancer with PD-L1 50% or more (EMPOWER-Lung 1): 35-month follow-up from a mutlicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2023 Sep;24(9):989-1001. doi: 10.1016/S1470-2045(23)00329-7. Epub 2023 Aug 14. PMID 37591293
- [Background] Hellmann MD, Paz-Ares L, Bernabe Caro R, Zurawski B, Kim SW, Carcereny Costa E, Park K, Alexandru A, Lupinacci L, de la Mora Jimenez E, Sakai H, Albert I, Vergnenegre A, Peters S, Syrigos K, Barlesi F, Reck M, Borghaei H, Brahmer JR, O'Byrne KJ, Geese WJ, Bhagavatheeswaran P, Rabindran SK, Kasinathan RS, Nathan FE, Ramalingam SS. Nivolumab plus Ipilimumab in Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2019 Nov 21;381(21):2020-2031. doi: 10.1056/NEJMoa1910231. Epub 2019 Sep 28. PMID 31562796
- [Background] Jakowlew SB. Transforming growth factor-beta in cancer and metastasis. Cancer Metastasis Rev. 2006 Sep;25(3):435-57. doi: 10.1007/s10555-006-9006-2. PMID 16951986
- [Background] Huber-Ruano I, Raventos C, Cuartas I, Sanchez-Jaro C, Arias A, Parra JL, Wosikowski K, Janicot M, Seoane J. An antisense oligonucleotide targeting TGF-beta2 inhibits lung metastasis and induces CD86 expression in tumor-associated macrophages. Ann Oncol. 2017 Sep 1;28(9):2278-2285. doi: 10.1093/annonc/mdx314. PMID 28911087
- [Background] Bierie B, Moses HL. Tumour microenvironment: TGFbeta: the molecular Jekyll and Hyde of cancer. Nat Rev Cancer. 2006 Jul;6(7):506-20. doi: 10.1038/nrc1926. PMID 16794634
- [Background] Tauriello DVF, Palomo-Ponce S, Stork D, Berenguer-Llergo A, Badia-Ramentol J, Iglesias M, Sevillano M, Ibiza S, Canellas A, Hernando-Momblona X, Byrom D, Matarin JA, Calon A, Rivas EI, Nebreda AR, Riera A, Attolini CS, Batlle E. TGFbeta drives immune evasion in genetically reconstituted colon cancer metastasis. Nature. 2018 Feb 22;554(7693):538-543. doi: 10.1038/nature25492. Epub 2018 Feb 14. PMID 29443964
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leal TA, Riess JW, Jensen E, Zhao B, Pietanza MC, Brahmer JR. Five-Year Outcomes With Pembrolizumab Versus Chemotherapy for Metastatic Non-Small-Cell Lung Cancer With PD-L1 Tumor Proportion Score >/= 50. J Clin Oncol. 2021 Jul 20;39(21):2339-2349. doi: 10.1200/JCO.21.00174. Epub 2021 Apr 19. PMID 33872070
- [Background] Uckun FM, Qazi S, Trieu VN. Proof of concept for the clinical utility of a convection enhanced delivery platform for immune-oncology drugs against brain tumors. Cancer Rep Rev. 2020;3:1-8
- [Background] Jaschinski F, Korhonen H, Janicot M. Design and Selection of Antisense Oligonucleotides Targeting Transforming Growth Factor Beta (TGF-beta) Isoform mRNAs for the Treatment of Solid Tumors. Methods Mol Biol. 2015;1317:137-51. doi: 10.1007/978-1-4939-2727-2_9. PMID 26072406
- [Background] Jaschinski F, Rothhammer T, Jachimczak P, Seitz C, Schneider A, Schlingensiepen KH. The antisense oligonucleotide trabedersen (AP 12009) for the targeted inhibition of TGF-beta2. Curr Pharm Biotechnol. 2011 Dec;12(12):2203-13. doi: 10.2174/138920111798808266. PMID 21619536
- [Background] Morris JC, Tan AR, Olencki TE, Shapiro GI, Dezube BJ, Reiss M, Hsu FJ, Berzofsky JA, Lawrence DP. Phase I study of GC1008 (fresolimumab): a human anti-transforming growth factor-beta (TGFbeta) monoclonal antibody in patients with advanced malignant melanoma or renal cell carcinoma. PLoS One. 2014 Mar 11;9(3):e90353. doi: 10.1371/journal.pone.0090353. eCollection 2014. PMID 24618589
- [Background] Serova M, Tijeras-Raballand A, Dos Santos C, Albuquerque M, Paradis V, Neuzillet C, Benhadji KA, Raymond E, Faivre S, de Gramont A. Effects of TGF-beta signalling inhibition with galunisertib (LY2157299) in hepatocellular carcinoma models and in ex vivo whole tumor tissue samples from patients. Oncotarget. 2015 Aug 28;6(25):21614-27. doi: 10.18632/oncotarget.4308. PMID 26057634
- [Background] Shull MM, Ormsby I, Kier AB, Pawlowski S, Diebold RJ, Yin M, Allen R, Sidman C, Proetzel G, Calvin D, et al. Targeted disruption of the mouse transforming growth factor-beta 1 gene results in multifocal inflammatory disease. Nature. 1992 Oct 22;359(6397):693-9. doi: 10.1038/359693a0. PMID 1436033
- [Background] Saika S, Saika S, Liu CY, Azhar M, Sanford LP, Doetschman T, Gendron RL, Kao CW, Kao WW. TGFbeta2 in corneal morphogenesis during mouse embryonic development. Dev Biol. 2001 Dec 15;240(2):419-32. doi: 10.1006/dbio.2001.0480. PMID 11784073
- [Background] Hau P, Jachimczak P, Schlingensiepen R, Schulmeyer F, Jauch T, Steinbrecher A, Brawanski A, Proescholdt M, Schlaier J, Buchroithner J, Pichler J, Wurm G, Mehdorn M, Strege R, Schuierer G, Villarrubia V, Fellner F, Jansen O, Straube T, Nohria V, Goldbrunner M, Kunst M, Schmaus S, Stauder G, Bogdahn U, Schlingensiepen KH. Inhibition of TGF-beta2 with AP 12009 in recurrent malignant gliomas: from preclinical to phase I/II studies. Oligonucleotides. 2007 Summer;17(2):201-12. doi: 10.1089/oli.2006.0053. PMID 17638524
- [Background] Bogdahn U, Hau P, Stockhammer G, Venkataramana NK, Mahapatra AK, Suri A, Balasubramaniam A, Nair S, Oliushine V, Parfenov V, Poverennova I, Zaaroor M, Jachimczak P, Ludwig S, Schmaus S, Heinrichs H, Schlingensiepen KH; Trabedersen Glioma Study Group. Targeted therapy for high-grade glioma with the TGF-beta2 inhibitor trabedersen: results of a randomized and controlled phase IIb study. Neuro Oncol. 2011 Jan;13(1):132-42. doi: 10.1093/neuonc/noq142. Epub 2010 Oct 27. PMID 20980335
- [Background] Mariathasan S, Turley SJ, Nickles D, Castiglioni A, Yuen K, Wang Y, Kadel EE III, Koeppen H, Astarita JL, Cubas R, Jhunjhunwala S, Banchereau R, Yang Y, Guan Y, Chalouni C, Ziai J, Senbabaoglu Y, Santoro S, Sheinson D, Hung J, Giltnane JM, Pierce AA, Mesh K, Lianoglou S, Riegler J, Carano RAD, Eriksson P, Hoglund M, Somarriba L, Halligan DL, van der Heijden MS, Loriot Y, Rosenberg JE, Fong L, Mellman I, Chen DS, Green M, Derleth C, Fine GD, Hegde PS, Bourgon R, Powles T. TGFbeta attenuates tumour response to PD-L1 blockade by contributing to exclusion of T cells. Nature. 2018 Feb 22;554(7693):544-548. doi: 10.1038/nature25501. Epub 2018 Feb 14. PMID 29443960
- [Background] Ganesh K, Massague J. TGF-beta Inhibition and Immunotherapy: Checkmate. Immunity. 2018 Apr 17;48(4):626-628. doi: 10.1016/j.immuni.2018.03.037. PMID 29669246
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Background] Trieu V, Wang W, Qazi S, et al. IL-8 as PD biomarker for TGF-b antisense (OT-101) therapy: Results of a phase II trial. Journal of Clinical Oncology 35, no. 15_suppl. DOI: 10.1200/JCO.2017.35.15_suppl.e15742
- [Background] D'Cruz OJ, Qazi S, Hwang L, Ng K, Trieu V. Impact of targeting transforming growth factor beta-2 with antisense OT-101 on the cytokine and chemokine profile in patients with advanced pancreatic cancer. Onco Targets Ther. 2018 May 14;11:2779-2796. doi: 10.2147/OTT.S161905. eCollection 2018. PMID 29785126
- [Background] Liu, S & Yuan, Y 2015, 'Bayesian optimal interval designs for phase I clinical trials', Journal of the Royal Statistical Society. Series C: Applied Statistics, vol. 64, no. 3, pp. 507-523. https://doi.org/10.1111/rssc.12089
- [Background] Yuan Y, Hess KR, Hilsenbeck SG, Gilbert MR. Bayesian Optimal Interval Design: A Simple and Well-Performing Design for Phase I Oncology Trials. Clin Cancer Res. 2016 Sep 1;22(17):4291-301. doi: 10.1158/1078-0432.CCR-16-0592. Epub 2016 Jul 12. PMID 27407096
- [Background] Zhou H, Yuan Y, Nie L. Accuracy, Safety, and Reliability of Novel Phase I Trial Designs. Clin Cancer Res. 2018 Sep 15;24(18):4357-4364. doi: 10.1158/1078-0432.CCR-18-0168. Epub 2018 Apr 16. PMID 29661774
- [Background] Venier J., Herrick R., Norris C., Liu S., Zhang L., Yuan Y., Lin R., & Zhou H. (2021). Bayesian Optimal Interval (BOIN) Phase I Design (PID-862): Version 1.1.0, Houston, Texas: The University of Texas MD Anderson Cancer Center Available at: https://biostatistics.mdanderson.org/SoftwareDownload/
- [Background] Ivanova A, Qaqish BF, Schell MJ. Continuous toxicity monitoring in phase II trials in oncology. Biometrics. 2005 Jun;61(2):540-5. doi: 10.1111/j.1541-0420.2005.00311.x. PMID 16011702
- See also: Pharmacokinetic-Pharmacodynamic (PKPD) Analysis For P001 - Phase 1/2 Clinical Trial For OT-101 Against Pancreatic Cancer, Melanoma, and Colorectal Cancer — https://www.oncotelic.com/wp-content/uploads/2022/07/JCA-2022.pptx.pdf
- See also: Mechanism of Action for OT-101 TGF-β Immunotherapy — https://www.oncotelic.com/wp-content/uploads/2022/11/ASCO-SITC-2022-Final-revised2.pdf